CLINICAL TRIAL: NCT02497339
Title: Mindfulness Training for Smoking Cessation in Women in the Workplace - a Pilot Randomized Controlled Trial
Brief Title: Mindfulness Training for Smoking Cessation in Women in Workplaces
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Lok Sin Tong Benevolent Society, Kowloon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: LSTWomen
Record Dates: First submitted 2015-07-09; First posted 2015-07-14 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation interventions; mindfulness training
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Intervention group (Experimental): Intervention group (Mindfulness Smoking cessation program): Women in intervention group will be provided 2 sessions mindfulness training within 2 weeks. Each session will last for 2 hours with 8-20 participants. For mindfulness training, it aims to understand women smokers' own life planning, stressors and their correlation with smoking; to help women smokers sit with negative affect and alleviate stress through mindfulness; to educate women smokers gain the self-control and replace the smoking habit; to teach women smokers how to prevent craving and relapse.
  Interventions: Behavioral: Mindfulness training
- Control group (Experimental): Control group (Self-help smoking cessation booklet): Only the self-help booklet related to quitting will be provided to the participants.
  Interventions: Behavioral: Mindfulness training

INTERVENTIONS:
Behavioral: Mindfulness training — Using mindfulness training (Thinking and Yoga class) to help women smokers in workplaces to quit smoking

SUMMARY:
This study has the following objectives:

1. To raise the awareness of female smokers about the harmfulness of tobacco towards their life issues
2. To encourage female smokers to stop using tobacco
3. To assess the effectiveness of mindfulness approach for smoking cessation in women

We will use cluster randomisation. About 40 companies (5 smokers / company) involved in the study will be matched on the company characteristics (e.g. company size, the industry the company belongs to). Using random generator in Excel, random number will be first generated to each pair i.e. there will be 1-40 random numbers. For each pair, the two companies will be randomly assigned to 0 or 1. Companies who are assigned to 1 will be allocated to intervention . Interviewers (assessors) in the follow-ups will not be involved in the randomization process and be totally blinded to the group assignment (allocation concealment).

Invitation letter will be sent to beauty and retail industries or other women-related industries by Lok Sin Tong. Health talks on smoking and its hazard will deliver to each company. For those who join the workshops after the health talks will fill in pre- and post- workshop questionnaires (Appendix 4-5). Women who attend the health talk will be recruited on site. Women will be screened by the criteria of eligibility form (Appendix 1) and all eligible women smokers will be asked to sign on informed consents (Appendix 2, 3) before they participate in the programs. After they consent to participate, they will fill in a baseline questionnaire (Appendix 6), and will be assigned to intervention or control group according to the allocation of their company. Some of the eligible women may miss the health talks and directly join the intervention program, because of this situation the intervention group will be further divided into Group A and B: women in Group A will attend health talks and intervention program, women in Group B will only attend intervention program.

Intervention group (Mindfulness Smoking cessation program): Women in intervention group will be provided 2 sessions mindfulness training within 2 weeks. Each session will last for 2 hours with 8-20 participants. For mindfulness training, it aims to understand women smokers' own life planning, stressors and their correlation with smoking; to help women smokers sit with negative affect and alleviate stress through mindfulness; to educate women smokers gain the self-control and replace the smoking habit; to teach women smokers how to prevent craving and relapse. The tentative agenda is shown below:

Session 1 (Introductory) Contents

1. Pre-questionnaire
2. Introducing mindfulness and managing craving with mindfulness
3. Understanding the components of craving and its management

   * The relationship between habitual response and learned association
   * The physiological and psychological withdrawal symptoms
4. Mindfulness yoga practices

Responsible person* Smoking Cessation Program in Workplace (SCPW) staff & Yoga teacher

Session 2 (Advanced)

Contents

1. Knowledge about impacts of smoking on women's health
2. Recapture the management of craving through mindfulness
3. Mindfulness exercises
4. Mindfulness yoga practices

Responsible person* SCPW staff & Yoga teacher

* SCPW staff would be responsible for the whole session except for the part "stress reduction and self-control through mindfulness yoga". It would be held by the yoga teacher.

Control group (Self-help smoking cessation booklet): Only the self-help booklet related to quitting will be provided to the participants.

Evaluation: 1-month telephone interviews will be conducted for control group at 1- (Appendix 97) and 6-month follow-ups will be conducted for both groups (after the last interventions) by trained interviewers (blinded to the group assignment). Participants who have reported abstinence in past 7 days from smoking at 6-month follow-ups will undergo a non-biochemical validation to check their quitting status. They will be invited to have biochemical validation tests (saliva cotinine test and exhaled CO test) at 6-month follow-up.

In-depth face-to-face interview will be conducted by trained interviewers in 10 randomly selected participants in each group (in total 20 participants) to better understand their quitting process, quitting difficulty, and their own feeling and experience in the project.

ELIGIBILITY:
Inclusion criteria:

* Women who smoked at least 1 cigarette a day by the time of the study starts
* Aged 18 or above
* Able to communicate in Cantonese or Mandarin, and read and write Chinese

Exclusion criteria:

* Women smokers with unstable physical or psychological conditions as advised by a doctor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Self-reported quit rate for the past 7 days | 6-month follow-up
  Quit rate of participants who stop smoking in the past 7 days

SECONDARY OUTCOMES:
Biochemically validated quit rate | 6-month follow-up
  Validated quit rate of participants who passed the bio-chemical validation for testing whether the participants have stopped smoking
50% smoking reduction | 6-month follow-up
  Reduce at least 50% cigarette consumption compared with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Man-ping Wang, PhD, Principal Investigator — School of Nursing, The University of Hong Kong
Locations (1):
- 2/F, 61 Lung Kong Rd, Kowloon City, Lok Sin Tong Benevolent Society, Hong Kong, China

REFERENCES:
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Jackson S, Brown J, Norris E, Livingstone-Banks J, Hayes E, Lindson N. Mindfulness for smoking cessation. Cochrane Database Syst Rev. 2022 Apr 14;4(4):CD013696. doi: 10.1002/14651858.CD013696.pub2. PMID 35420700